CLINICAL TRIAL: NCT00419497
Title: Paleolithic Diet in the Treatment of Glucose Intolerance
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lund University Hospital (Other)
Responsible Party: Principal Investigator, Staffan Lindeberg, Ass prof, Lund University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LU 665-02
Record Dates: First submitted 2007-01-04; First posted 2007-01-08 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Hyperglycemia; Coronary Heart Disease
Keywords: Paleolithic diet; Mediterranean-style diet; Glucose tolerance; Diabetes type 2; Weight loss; Waist
MeSH Terms: conditions — Hyperglycemia; Coronary Disease; Diabetes Mellitus, Type 2; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paleolithic diet vs Mediterranean diet (Active Comparator): Prudent diets with or without grains and dairy
  Interventions: Behavioral: Paleolithic diet vs Mediterranean diet

INTERVENTIONS:
Behavioral: Paleolithic diet vs Mediterranean diet — Prudent diets with or without grains and dairy

SUMMARY:
The purpose of this study is to determine whether a paleolithic diet improves glucose tolerance and insulin sensitivity in people with coronary heart disease and impaired glucose tolerance.

DETAILED DESCRIPTION:
There is uncertainty about the optimal diet in the prevention and treatment of glucose intolerance and diabetes type 2, disorders which are very common in patients with coronary heart disease (CHD). Earlier studies have generally focused on intakes of fat, carbohydrate, fiber, fruit and vegetables. Another approach compares foods that were available during human evolution with more recently introduced ones. Twenty-nine CHD patients with glucose intolerance or diabetes have been randomized to 1) a Paleolithic ("Old Stone Age") diet (n=14) based on lean meat, fish, fruit, vegetables, root vegetables, eggs, and nuts, or 2) a Consensus (Mediterranean-like) diet (n=15) based on whole grains, low-fat dairy products, vegetables, fruit, fish, and oils and margarines generally assumed to be healthy. Primary outcome variables are changes during 12 weeks in weight, waist circumference, and area under the curve for glucose (AUC Glucose0-120) and insulin (AUC Insulin0-120) at the oral glucose tolerance test.

ELIGIBILITY:
Inclusion Criteria:

* Hyperglycemia
* Coronary Heart Disease
* Increased waist circumference

Exclusion Criteria:

* Body mass index <20 kg/m2
* Serum creatinine >130 µmol/L
* Poor general condition
* Dementia
* Unwillingness/inability to prepare food at home (by study participant or partner)
* Participation in another medical trial
* Chronic inflammatory bowel disease
* Drug treatment with hypoglycemic agents
* Drug treatment with warfarin
* Drug treatment with oral steroid

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2003-01; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
change in weight and waist circumference | 12 weeks
area under the curve for glucose (AUC Glucose0-120) at the oral glucose tolerance test | 12 weeks
area under the curve for insulin (AUC Insulin0-120) at the oral glucose tolerance test | 12 weeks

SECONDARY OUTCOMES:
fasting plasma glucose | 12 weeks
30-min plasma glucose | 12 weeks
120-min plasma glucose | 12 weeks
fasting plasma insulin | 12 weeks
30-min plasma insulin | 12 weeks
120-min plasma insulin | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Staffan Lindeberg, MD PhD, Principal Investigator — Department of Clinical Sciences, IKVL 1, Lund University, Lund Sweden
Locations (1):
- Lund University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lindeberg S, Jonsson T, Granfeldt Y, Borgstrand E, Soffman J, Sjostrom K, Ahren B. A Palaeolithic diet improves glucose tolerance more than a Mediterranean-like diet in individuals with ischaemic heart disease. Diabetologia. 2007 Sep;50(9):1795-1807. doi: 10.1007/s00125-007-0716-y. Epub 2007 Jun 22. PMID 17583796
- [Derived] Jonsson T, Granfeldt Y, Erlanson-Albertsson C, Ahren B, Lindeberg S. A paleolithic diet is more satiating per calorie than a mediterranean-like diet in individuals with ischemic heart disease. Nutr Metab (Lond). 2010 Nov 30;7:85. doi: 10.1186/1743-7075-7-85. PMID 21118562